CLINICAL TRIAL: NCT01338493
Title: Maverick Total Disc Replacement in a 'Real World' Patient Population - A Prospective, Multicenter, Observational Study
Brief Title: Maverick Total Disc Replacement in a 'Real World' Patient Population
Acronym: Maverick
Status: Completed | Type: Observational
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Other Study IDs: Maverick Global Registry
Record Dates: First submitted 2011-02-17; First posted 2011-04-19 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lumbar spinal arthroplasty + Maverick™: Patients requiring total disc replacement
  Interventions: Procedure: lumbar spinal arthroplasty + Maverick™

INTERVENTIONS:
Procedure: lumbar spinal arthroplasty + Maverick™ — All patients will be subjected to a lumbar spinal arthroplasty. The anterior lumbar spine is approached through either a transperitoneal or retroperitoneal exposure. A complete anterior discectomy is performed and the Maverick™ Artificial Disc System is inserted to replace the damaged lumbar intervertebral disc.

SUMMARY:
The primary purpose of the study is to document the reduction of disability after Maverick total disc replacement surgery in a 'real-world' patient population requiring disc replacement.

ELIGIBILITY:
Inclusion criteria:

* Degenerative Disc Disease (DDD) defined as back pain of discogenic origin with degeneration of the disc confirmed by history and radiographic studies
* Foraminal stenosis due to loss of disc height
* Back pain and/or leg pain.

Exclusion criteria:

* Spondylolisthesis at the affected or adjacent level
* Posterior facet joint damage and/or disease at the affected level, including facet osteoarthritis, pars fracture and prior laminectomy
* Obesity
* Osteoporosis
* Metallic allergy to cobalt-chromium-molybdenum alloys
* Psychosis
* Infection
* Spinal canal stenosis
* Overlying thoracolumbar kyphosis
* Systemic infection or infection at the site of surgery
* Osteopenia, osteoporosis, or osteomalacia to a degree that spinal instrumentation would be contraindicated
* Diseases of bone metabolism
* Pregnancy
* Signs of local inflammation
* Fever or Leukocytosis
* Grossly distorted anatomy caused by congenital abnormalities
* Any other medical or surgical condition which would preclude the potential benefit of spinal implant surgery, such as the presence of congenital abnormalities, elevation of sedimentation rate unexplained by other diseases, elevation of white blood count (WBC), or a marked left shift in the WBC differential count (this also includes: spinal active oncology pathology; not healed fracture at treated or adjacent level)
* Any case where the implants or components selected would be too large or too small to achieve a successful result
* Any patient in which implant utilization would interfere with anatomical structures or expected physiological performance
* Any patient unwilling to follow postoperative instructions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient eligibility is determined according to labeling
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2009-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Le Huec, Prof., Principal Investigator — CHU Pellegrin Tripode
Locations (13):
- Montreal General Hospital, Québec, Canada
- France (9):
  - CHU Pellegrin Tripode, Bordeaux
  - CH Antoine Béclère - Service de Chirurgie Orthopédique, Clamart
  - Service de Chirurgie Orthopédique, AP-HP, Hôpital Beaujon, Clichy
  - Clinique de Neurochirurgie Hôpital Roger Salengro, Lille
  - CH La Timone, Marseille
  - CH de Meulan - Service de Chirurgie Orthopédique, Meulan-en-Yvelines
  - Service de Neurochirurgie Hôpital Nice, Nice
  - CH Lariboisière, Service de Neurochirurgie, Paris
  - Clinique du Cours Dillon, Toulouse
- Germany (3):
  - Charité Berlin - Klinik für Orthopädie, Berlin
  - Universitätsklinikum Magdeburg, Magdeburg
  - Praxis für Orthopädie und Neurochirurgie Potsdam, Potsdam

RESULTS

PARTICIPANT FLOW:
Period: Enrolled
Arm/Group | Lumbar Spinal Arthroplasty + Maverick™
Started | 139
Completed | 134
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Patient not implanted | 4
Period: Implant
Arm/Group | Lumbar Spinal Arthroplasty + Maverick™
Started | 134
Completed | 134
Not Completed | 0
Period: Discharge
Arm/Group | Lumbar Spinal Arthroplasty + Maverick™
Started | 134
Completed | 132
Not Completed | 2
Not completed — Death | 1
Not completed — Missed visit | 1
Period: 6 Months Follow up
Arm/Group | Lumbar Spinal Arthroplasty + Maverick™
Started | 132
Completed | 113
Not Completed | 19
Not completed — Lost to Follow-up | 11
Not completed — Missed visit | 8
Period: 12 Months Follow up
Arm/Group | Lumbar Spinal Arthroplasty + Maverick™
Started | 113
Completed | 104
Not Completed | 9
Not completed — Lost to Follow-up | 9
Period: 24 Months Follow up
Arm/Group | Lumbar Spinal Arthroplasty + Maverick™
Started | 104
Completed | 104
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lumbar Spinal Arthroplasty + Maverick™
Number analyzed (Participants) | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 64
Region of Enrollment [Number; unit: participants]
  France | 79
  Canada | 5
  Germany | 50

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Disability at 6 Months Versus Baseline Using the Oswestry Disability Index (ODI)
Description: The Oswestry Disability Index (ODI) derives from the Oswestry Low Back Pain Questionnaire, it is used to measure disability for low back pain. The index is scored from 0 to 100; 0 meaning 'no disability' and 100 meaning 'maximum disability'.
Time Frame: 6 months
Population: Reduction of disability was calculated for patients having available data at both baseline and 6 months.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lumbar Spinal Arthroplasty + Maverick™
Number analyzed (Participants) | 122
units on a scale | -25.4 [-29.0 to -21.9]
Statistical Analysis 1: Comparison: Lumbar Spinal Arthroplasty + Maverick™; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Relief of Back Pain at 6 Months Versus Baseline Using the Back Pain Intensity Score Assessed on a 10 cm Visual Analogue Scale (VAS)
Description: Back Pain was documented in a Visual Analogue Scale where the patients marked the location on the 10-centimeter line corresponding to the amount of pain they experienced.
  0 = no pain, 10 = worst possible pain
Time Frame: 6 months
Population: Reduction of disability was calculated for patients having available data at both baseline and 6 months.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lumbar Spinal Arthroplasty + Maverick™
Number analyzed (Participants) | 108
units on a scale | -4.0 [-4.5 to -3.4]
Statistical Analysis 1: Comparison: Lumbar Spinal Arthroplasty + Maverick™; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 24 months
Description: Seriousness of AEs was not assessed when the data were collected so it is not possible to separate SAEs and Other (Non-serious) AEs for the Maverick Registry. The study is now closed and it would not be possible to go back to the sites to ask them to classify the AEs. All events are here-reported as SAEs.
Arm/Group | Lumbar Spinal Arthroplasty + Maverick™
Serious Adverse Events (participants affected / at risk) | 57/134
Other Adverse Events (participants affected / at risk) | 0/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumbar Spinal Arthroplasty + Maverick™ (N=134)
Abdominal wall related (General disorders) | 9 (9)
Neurologic - Access-related (Nervous system disorders) | 12 (13)
Neurologic - Late radiculopathy (not access-related) (Nervous system disorders) | 12 (13)
Vascular (Vascular disorders) | 3 (3)
Visceral - Bowel or Peritoneum (General disorders) | 1 (1)
Visceral - Genito-Urinary tract (General disorders) | 5 (5)
Subsidence / Impaction (Musculoskeletal and connective tissue disorders) | 1 (1)
Early non-specific low BP (General disorders) | 5 (5)
Late non-specific low BP (General disorders) | 6 (6)
Foreign body reaction (Immune system disorders) | 1 (1)
Other events (General disorders) | 24 (27)

LIMITATIONS AND CAVEATS:
Seriousness of AEs was not assessed when the data were collected so it is not possible to separate SAEs and Other (Non-serious) AEs for the Maverick Registry. All events are here-reported as SAEs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidential Information shall not be disclosed and shall be property of sponsor during the term of the agreement and for 3 years after agreement termination. Results might be published or presented, however sponsor should receive publication for review at least 90 days prior to submittal. Sponsor shall limit its review to a determination of whether Confidential Information is disclosed, to allow sponsor to protect its rights in copyrightable material, and to check for technical correctness.